CLINICAL TRIAL: NCT05619341
Title: Effect of Rate Of Delivery on Colonic Fermentation of inuliN (EON)
Acronym: EON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Robin Spiller, Professor of Gastroenterology, University of Nottingham
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: FMHS 17-0622
Record Dates: First submitted 2022-11-01; First posted 2022-11-16 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Irritable Bowel
Keywords: fermentation; gas; colonic; inulin; psyllium
MeSH Terms: conditions — Irritable Bowel Syndrome; Mucopolysaccharidosis IV | interventions — Psyllium; Inulin

STUDY DESIGN:
Intervention Model Description: 3 way cross-over
Who Masked: Participant
Masking Description: psyllium / maltodextrin added to 500ml water + inulin 20g
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- inulin (Placebo Comparator): 20g inulin in 500ml water
  Interventions: Dietary Supplement: inulin
- inulin + psyllium (Active Comparator): Inulin 20g + 20g psyllium in 500 ml water
  Interventions: Dietary Supplement: psyllium; Dietary Supplement: inulin
- inulin divided doses (Active Comparator): 2.5 g inulin in 62.5ml water given at 45 minute intervals
  Interventions: Dietary Supplement: inulin

INTERVENTIONS:
Dietary Supplement: psyllium — psyllium 20g
  Arms: inulin + psyllium
Dietary Supplement: inulin — long chain fructan

SUMMARY:
To test whether slowing the rate of delivery of inulin with either psyllium or divided dosing of inulin, will reduce colonic gas production as compared to inulin combined with placebo.

To obtain pilot data on link between habitual diet and fermentation of inulin.

DETAILED DESCRIPTION:
Our challenge is to understand how fibre interacts with whole-gut function to alter colonic fermentation of fermentable oligo-di-mono-saccharides and polyhydric alcohols (FODMAPs). We have previously performed the study entitled the Effect of modified Cellulose On COlonic fermentAtion of inulin (COCOA) in which a modified methylcellulose (food grade product -modified celluloses- which can form gels at body temperature ) was used and showed some reduction, but this was not statistically significant, and much less than with psyllium. We wish to determine whether slowing delivery of inulin will produce a lowering of breath hydrogen equivalent to that seen with psyllium. We also found that the breath hydrogen curve had not shown a consistent fall by 6 hours suggesting that 6 hours was not long enough to accurately define the area under the curve (AUC). We now plan to use breath sampling bags to collect breath samples at home to define the breath hydrogen response over whole 24-hour period post ingestion of test drink. We also hypothesise that the colonic microbiota will influence the fermentation of inulin and will collect stool samples to allow future work to correlate microbiota with fermentation rates as part of a separate Medical Research Council funded study.

Aim Our aim is to test the hypothesis that slowing delivery of inulin will achieve a similar reduction in breath hydrogen production over the 24 hours following ingestion as seen when co-administered with psyllium.

Objective The primary objective is to compare the effect of bolus administration of inulin (co-administrated with psyllium or maltodextrin placebo) with divided dose delivery of inulin over 6 hours on total gas production over 24 hours.

Secondary Objectives Secondary objectives will be 1) to compare breath hydrogen AUC 0-24h with values based on AUC 0-6h that was assessed in the previous study (COCOA) to see how much the shorter period underestimates H2 production; 2) to assess breath methane production AUC 0-24h after consumption of test drinks; and 3) to collect pilot data on habitual dietary FODMAPs intake to assess whether this alters fermentation of inulin.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older.
* Able to give informed consent.
* Scoring ≤3 (i.e., mild, or less) for symptoms of flatulence, bloating and abdominal pain in previous 2 weeks using a modified Gastrointestinal Symptom Rating Scale (5).
* Agrees to consume the meals provided.
* Agrees to not smoke during the breath hydrogen sampling period

Exclusion Criteria:

* Pregnancy declared by candidate.
* History declared by the candidate of pre-existing gastrointestinal disorder that may affect bowel function.
* Reported history of previous resection of the oesophagus, stomach, or intestine (excluding appendix).
* Intestinal stoma.
* Any medical condition potentially compromising participation in the study e.g., type 1 diabetes mellitus, respiratory disease limiting ability to use breath hydrogen analyser, known intolerance to one of the test substances.
* Will not agree to dietary restrictions required nor consume the standard meals required during the study day.
* Unable to stop drugs known to alter GI motility including mebeverine, opiates, monoamine oxidase inhibitors, phenothiazines, benzodiazepines, calcium channel antagonists for the duration of the study (Selective serotonin reuptake inhibitors, low dose tricyclic antidepressants, antihistamines, and oral contraceptive pill will be recorded in the CRF but will not be an exclusion criteria).
* Participants who are taking antibiotics or probiotics as they might alter gut microbiota.
* Poor understanding of English language.
* Participation in night shift work the week prior to the study day. Night work is defined as working between midnight and 6.00 AM.
* Anyone who in the opinion of the investigator is unlikely to be able to comply with the protocol e.g., cognitive dysfunction, chaotic lifestyle related to substance abuse.
* Having taken part in a research study in the last 3 months involving invasive procedures or an inconvenience allowance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Hydrogen production | 2 days
  AUC 0-24h

SECONDARY OUTCOMES:
Methane production | 2 days
  AUC 0-24h
Intake of FOOMDAPS | 4 days
  24 h food diary X 4

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham Digestive Disease Centre, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Galvin MA, Kiely M, Harrington KE, Robson PJ, Moore R, Flynn A. The North/South Ireland Food Consumption Survey: the dietary fibre intake of Irish adults. Public Health Nutr. 2001 Oct;4(5A):1061-8. doi: 10.1079/phn2001187. PMID 11820919
- [Result] Dionne J, Ford AC, Yuan Y, Chey WD, Lacy BE, Saito YA, Quigley EMM, Moayyedi P. A Systematic Review and Meta-Analysis Evaluating the Efficacy of a Gluten-Free Diet and a Low FODMAPs Diet in Treating Symptoms of Irritable Bowel Syndrome. Am J Gastroenterol. 2018 Sep;113(9):1290-1300. doi: 10.1038/s41395-018-0195-4. Epub 2018 Jul 26. PMID 30046155
- [Result] Gunn D, Abbas Z, Harris HC, Major G, Hoad C, Gowland P, Marciani L, Gill SK, Warren FJ, Rossi M, Remes-Troche JM, Whelan K, Spiller RC. Psyllium reduces inulin-induced colonic gas production in IBS: MRI and in vitro fermentation studies. Gut. 2022 May;71(5):919-927. doi: 10.1136/gutjnl-2021-324784. Epub 2021 Aug 5. PMID 34353864
- [Derived] Alhasani AT, Modasia AA, Anodiyil M, Corsetti M, Aliyu AI, Crooks C, Marciani L, Reid J, Yakubov GE, Taylor M, Avery A, Harris H, Warren FJ, Spiller RC. Mode of Action of Psyllium in Reducing Gas Production from Inulin and its Interaction with Colonic Microbiota: A 24-hour, Randomized, Placebo-Controlled Trial in Healthy Human Volunteers. J Nutr. 2025 Mar;155(3):839-848. doi: 10.1016/j.tjnut.2024.12.017. Epub 2024 Dec 26. PMID 39732438